CLINICAL TRIAL: NCT04939012
Title: Implementation of a Patient-centered, Reproductive Planning Decision Support Tool (MyPath) Among Women With Substance Use Disorder in the Immediate Postpartum Period
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Krans, MD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20110324; 1R01DA051674-01A1 (NIH)
Record Dates: First submitted 2021-06-23; First posted 2021-06-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Substance Use Disorders; Pregnancy Related; Contraception
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyPath Intervention (Experimental): At the first visit participants randomized to this arm receive MyPath contraceptive decision tool.
  Interventions: Behavioral: MyPath Intervention
- Standard of Care (Active Comparator): At the first visit participants randomized to this arm receive standard of care contraceptive counseling.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: MyPath Intervention — MyPath is a novel patient-centered, reproductive planning decision support tool developed by the research team used to facilitate postpartum contraceptive decision-making among women with SUDs. Designed to facilitate high-quality decisions regarding pregnancy and contraception, MyPath helps women a) review their thoughts about pregnancy and children, b) learn about fertility and preconception health and c) prioritize their preferences for various contraceptive method characteristics (e.g. effectiveness, side effects). As such, MyPath uses a patient-centered approach to help women frame their contraceptive decisions in the context of their goals and health and is a critical first step towards addressing reproductive health inequities among women with SUDs.
  Arms: MyPath Intervention
Behavioral: Usual care — Standard of Care
  Arms: Standard of Care

SUMMARY:
This is a study to determine the effect of a novel patient-centered, reproductive planning decision support tool developed by the research team called MyPath on postpartum contraceptive decision-making among women with SUDs.

DETAILED DESCRIPTION:
The reproductive health needs of women with substance use disorders (SUDs) are unmet. Over 80% of pregnancies among women with SUDs are unintended, compared to 45% of the general population, and over 20% of women with SUDs have had a short interpregnancy interval (i.e. ≤ 18 months after a previous birth). Adverse reproductive health outcomes are perpetuated by contraceptive decisions that are inconsistent with women's reproductive goals. In an evaluation of women in opioid use disorder (OUD) treatment, only half of sexually active women not wanting to get pregnant used contraception, with condoms the most frequent method used. Pregnancy is a unique opportunity to address contraceptive needs due to increased healthcare access and expanded Medicaid eligibility, increased access to highly effective methods such as long-acting reversible contraception (LARC) and enhanced motivation to avoid rapid, repeat pregnancy. Despite this, over 75% of women with OUD do not use postpartum contraception and less than 2% receive LARC.

Currently, there are no effective strategies to improve postpartum contraceptive decision-making for women with SUDs. As an initial step to address this gap, the investigators conducted an observational study of postpartum contraceptive choices among 194 women with OUD at our maternity hospital (Plan NOW). Per usual care, women were provided with information about all contraceptive options, consistent with "information-based" counseling, and access to all methods including immediate postpartum LARC. Several findings informed this proposal. First, women's postpartum contraceptive decisions were often inconsistent with their childbearing goals. Among women who did not want another child, 36% did not choose a highly effective method and 10% had a repeat pregnancy within one year. Second, women had limited contraceptive knowledge and frequent misconceptions about their fertility and vulnerability to pregnancy. Third, women's decisional autonomy regarding sex and contraception was often threatened due to ongoing illicit drug use and reproductive coercion by partners. Fourth, women who wanted another baby did not feel supported and often felt pressured to choose a highly effective method. Therefore, failure to frame contraceptive decisions within the larger reproductive health context of women with OUD was a major barrier to high quality decision-making.

The goal of this research is to help women with SUDs make informed decisions about their reproductive health that align with their preferences, values and reproductive goals. Our objective in this application is to determine the effect of a novel patient-centered, reproductive planning decision support tool developed by the research team called MyPath on postpartum contraceptive decision-making among women with SUDs. Designed to facilitate high-quality decisions regarding pregnancy and contraception, MyPath helps women a) review their thoughts about pregnancy and children, b) learn about fertility and preconception health and c) prioritize their preferences for various contraceptive method characteristics (e.g. effectiveness, side effects). As such, MyPath uses a patient-centered approach to help women frame their contraceptive decisions in the context of their goals and health and is a critical first step towards addressing reproductive health inequities among women with SUDs. Our overarching hypothesis is that patient-centered, reproductive planning decision support will facilitate high quality decision-making and thus improve postpartum contraceptive utilization and reproductive health outcomes among women with SUDs. To test this hypothesis, the investigators propose a hybrid type 1 effectiveness-implementation randomized controlled trial, guided by the following aims:

Aim 1: Assess the effect of patient-centered, reproductive planning decision support (MyPath) on postpartum contraceptive utilization and reproductive health outcomes among women with SUDs

Aim 2: Determine if the relationship between MyPath and contraceptive utilization is mediated by decision quality. Decision quality will be measured using four patient-centered components of decision-making: knowledge, values concordance, decisional conflict and involvement. The investigators hypothesize that improvements in decision quality will mediate the relationship between MyPath and contraceptive utilization.

Aim 3: Identify barriers and facilitators to integrating MyPath into routine postpartum clinical care. The investigators will gather process evaluation data during the randomized controlled trial (RCT) and conduct qualitative interviews with key patient, provider and health system stakeholders to identify potential barriers and facilitators to future implementation in maternity settings and routine postpartum clinical care, if MyPath is found to be effective.

ELIGIBILITY:
Inclusion Criteria

Prenatal Cohort:

* Be greater than or equal to 18 years of age.
* Be pregnant with an EGA of 22 to 37 weeks at enrollment.
* Plan to deliver at MWH.
* Meet DSM-5 criteria for a SUD (i.e., opioid, stimulant or other use disorder) and/or have a diagnosis code for a substance use disorder in their medical record.

Postpartum Cohort:

* Be greater than or equal to 18 years of age.
* Be 0-9 days postpartum at enrollment.
* Have delivered at MWH.
* Meet DSM-5 criteria for a SUD (i.e., opioid, stimulant or other use disorder) and/or have a diagnosis code for a substance use disorder in their medical record.

Exclusion Criteria:

* Have had a fetal or neonatal death with their current pregnancy.
* Be currently in jail or prison as required by court of law. Persons on probation or in residential facilities do not need to be excluded.
* Have any other condition (social or medical) which, in the opinion of the Investigator, would make study participation unsafe, make study participation difficult, and/or complicate data interpretation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Contraceptive method continuation | Delivery (Immediate Post-delivery Inpatient Visit) to 18 months post delivery
  Contraceptive method continuation as measured at each postpartum follow-up assessment by participants use of the same contraceptive method as she did at the previous timepoint.
Continuous contraceptive use | Delivery (Immediate Post-delivery Inpatient Visit) to 18 months post delivery
  Continuous contraceptive use as measured by participants continuously using any moderately (i.e., pill, patch, or ring, injection) or highly effective (i.e., long-acting reversible contraceptive (LARC), tubal ligation) method at consecutive timepoints. Reasons for stopping or switching methods will also be obtained.

SECONDARY OUTCOMES:
Use of moderate or highly effective method | Delivery (Immediate Post-delivery Inpatient Visit) to 18 months post delivery
  Use of moderate or highly effective method as measured by participants who select any moderately (i.e., pill, patch, or ring, injection) or highly effective (i.e., long-acting reversible contraceptive (LARC), tubal ligation) method at any timepoint.
Unintended pregnancy | Delivery (Immediate Post-delivery Inpatient Visit) to 18 months post delivery
  Rate of unintentional pregnancy as measured by number of women having a new pregnancy, evaluation of intendedness of that pregnancy with the 6-item London Measure of Unplanned Pregnancy (LMUP).
Interpregnancy interval | Delivery (Immediate Post-delivery Inpatient Visit) to 18 months post delivery
  Time-to-next pregnancy as measured by time-to-event analyses.
Decisional Conflict | Enrollment (22 - 37 weeks pregnant) to 18 months post delivery
  Decisional conflict as measured by the Decision Conflict Scale (DCS).
Values concordance | Enrollment (22 - 37 weeks pregnant) to 18 months post delivery
  We will measure women's perceptions of the values concordance of their selected postpartum contraceptive method as measured by a two-item adapted Measure of the Alignment of Choices (MATCH)
Knowledge | Enrollment (22 - 37 weeks pregnant) to 18 months post delivery
  Reproductive planning knowledge as measured by an 18-item reproductive planning knowledge scale adapted from validated contraceptive knowledge assessments.
Involvement | Enrollment (22 - 37 weeks pregnant) to 18 months post delivery
  Involvement in decision making as measured by the Interpersonal Quality in Family Planning care (IQFP).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Krans, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share data acquired through this study, however the research team may share de-identified data in the future.